CLINICAL TRIAL: NCT01851941
Title: A Phase II Trial of Perioperative Chemotherapy With Oxaliplatin, 5-Fluorouracil, Leucovorin(MODIFIED FOLFOX6) in Patients With Locally Advanced Operable Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seock-Ah Im, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H 0406127 007; H 0406127 007 (Other: Seoul National University Hospital)
Record Dates: First submitted 2013-05-06; First posted 2013-05-13 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Advanced Gastric Cancer
MeSH Terms: interventions — Leucovorin; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mFOLFOX6 (Experimental): Modified FOLFOX6 regimen consists of oxaliplatin 100 mg/m2 and FA 100 mg/m2 given as a 2 hour intravenous infusion, followed by 5-FU 2.4 g/m2 given as a continuous infusion over 46 hour, which is repeated every 2 weeks. Patients receive 4 cycles of neoadjuvant modified FOLFOX6 followed by curative radical surgery with D2 dissection and 4 cycles of adjuvant modified FOLFOX6.
  Interventions: Drug: mFOLFOX6 (folinic acid, 5-fluorouracil, and oxaliplatin )

INTERVENTIONS:
Drug: mFOLFOX6 (folinic acid, 5-fluorouracil, and oxaliplatin ) — Modified FOLFOX6 regimen consists of oxaliplatin 100 mg/m2 and FA 100 mg/m2 given as a 2 hour intravenous infusion, followed by 5-FU 2.4 g/m2 given as a continuous infusion over 46 hour, which is repeated every 2 weeks. Patients receive 4 cycles of neoadjuvant modified FOLFOX6 followed by curative radical surgery with D2 dissection and 4 cycles of adjuvant modified FOLFOX6.

SUMMARY:
The role of perioperative chemotherapy in potentially operable advanced gastric cancer (AGC) with regional lymph node metastasis is still in the area of controversy. The aim of this study is to evaluate the efficacy and toxicity of folinic acid (FA), infusional 5-fluorouracil (5-FU), and oxaliplatin (modified FOLFOX6) in potentially resectable AGC with regional lymph node (LN) metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated patients with pathologically proven advanced gastric adenocarcinoma with regional LN metastasis (clinical stage: cT2-4 and N+)
* At least one measurable regional lymph node metastasis according to the Response Evaluation Criteria in Solid Tumors (RECIST v. 1.0)
* age between 18 and 75 years
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1
* no prior chemotherapy or radiotherapy
* adequate bone marrow, hepatic and renal function (absolute neutrophil count [ANC] ≥ 1.5ⅹ109/L, platelet count ≥ 100ⅹ109/L, total bilirubin ≤ 1.5ⅹupper limit of normal [ULN], serum transaminases ≤ 2.5ⅹULN, alkaline phosphatase ≤ 2.5ⅹULN, serum creatinine ≤ 1.5ⅹULN or actual or calculated creatinine clearance ≥ 50 mL/min).

Exclusion Criteria:

* clinical stage T1 tumors
* clinical or radiologic evidence of distant metastasis
* intestinal obstruction or impending obstruction
* active tumor bleeding
* interstitial pneumonitis or symptomatic pulmonary fibrosis
* peripheral neuropathy of National Cancer Institute Common Toxicity Criteria (NCI-CTC) grade ≥1
* pregnant or breastfeeding patients
* other serious diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2004-10; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
clinical response rate as assessed using RECIST criteria, with computed tomography (CT) scans at baseline and after 4cycles of chemotherapy | 4 cycles of chemotherapy (expected average of 8 weeks)

SECONDARY OUTCOMES:
Time to progression | From date of study enrollment until the date of first documented progression, assessed up to 60 months
overall survival | From date of study enrollment until the date of first documented progression, assessed up to 60 months

OTHER OUTCOMES:
gene expression profile | after 4 cycles of chemotherapy (expected average of 8 weeks)
early metabolic response by PET-CT | 2 cycles of chemotherapy (expected average of 4 weeks)
Pharmacologic Genetic Marker | 4 cycles of chemotherapy (expected average of 8 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea